CLINICAL TRIAL: NCT01440894
Title: Verify the Functions and Efficiency of Transtek Glass Body Fat Analyzer, GBF-733-W1, GBF-1012, BF-1039, BF-1041-A, GBF-950-D.
Brief Title: Clinical Trail of Transtek Glass Body Fat Analyzer
Acronym: GBFA
Status: Completed | Type: Observational
Sponsor: Leo Wang (Other)
Collaborators: BTS International (Other)
Responsible Party: Sponsor-Investigator, Leo Wang, Team leader, BTS International
Organization: BTS International (Other)
Other Study IDs: TranstekGBFA11003; BTS-TRANS03 (Other: BTSInternational)
Record Dates: First submitted 2011-09-25; First posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Weight; Body Fat Disorder; Bone Mass
Keywords: weight; body fat; total body water; bone mass; muscle mass
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Body Analysis
  Interventions: Device: Comparison test

INTERVENTIONS:
Device: Comparison test — Reference Device: Transtek Glass Body Analyzer, GBF-950, accuracy: ±0.1kg and range: 0-180kg.
  DUT(Device Under Test): Transtek Glass Body Fat Analyzer, Model: GBF-733-W1, GBF-1012, BF-1039, BF-1041-A, and GBF-950-D.
  Other Names: Brand name: Transtek

SUMMARY:
The clinical protocol of the clinical testing of this device:

1. Objective of the test: To verify the functions and efficiency of devices.
2. Test methods and procedures: Comparison Test.
3. DUT(Device Under Test): Transtek Glass Body Fat Analyzer, Model: GBF-733-W1, GBF-1012, BF-1039, BF-1041-A, and GBF-950-D.
4. Comparison device: Transtek Glass Body Analyzer, GBF-950 (Predicate Device).
5. Study endpoints: Transtek devices and the predicate device are substantial equivalence.
6. Statistical methodology used: Description of statistical methods.
7. Result: Efficiencies of Transtek devices and predicate device are in the same level.

DETAILED DESCRIPTION:
Hospital Information The data was collected by Zhongshan City People's Hospital Clinical Investigator Team at Zhongshan City People's Hospital, No.2 Sunwen Dong Road, Zhongshan, Guangdong 528403, P. R. China.

Investigator: Dr. Stephen Feng, Leader; Fan Futao, Nurse A; Wu Yanting, Nurse B.

Contact Dr. James Zhu Tel: +86 760 88823818 Used Equipments DUT (Device Under Test): Transtek Glass Body Fat Analyzer, Model: GBF-733-W1, GBF-1012, BF-1039, BF-1041-A, and GBF-950-D.

Reference Device: Transtek Glass Body Analyzer, GBF-950 (Predicate Device). Test Protocol

1. Test Purpose:

   The aim of clinical test is to collect weight, body fat, total body water, bone mass, and muscle mass reading value which measured by DUT and reference device.

   Note: GBF-733-W1 and BF-1039 have not bone mass functions. So it just collects weight, body fat, total body water, and muscle mass data.
2. Target Subject:

   The subject database shall contain at least 25 male and 25 female subjects and all above 18 years old. Patient's population analysis is bellow.
3. Test procedures 1) Record the name, age, and gender values of each subject. 2) Let subject seated calmly for two minutes before test, dry the feet. 3) Use device to measure weight, body fat, total body water, bone mass, and muscle mass; record reading value.

4) For each subject, repeat 3) to get 3 pairs measurements. 5) Repeat step 1) to 4) for every device (DUT: GBF-733-W1, GBF-1012, BF-1039, BF-1041-A, and GBF-950-D; and reference device: GBF-950).

6) Repeat step 1) to 5) for each subject. 5. Note:

1. No motion and speaking are allowed during the measurement.
2. All DUT use the same algorithms, have the same number of electrodes and contact the patient at the same body locations (feet), and operate on the same frequency.
3. Test environment: Temperature: 22±1℃; Relative humidity: 40~50%.

ELIGIBILITY:
Inclusion Criteria:

* male,female

Exclusion Criteria:

* below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population included patients whose age is above 18 years old. Male or Female.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Verify the accuracy of measure functions of device | 8 days
  Verify the functions and efficiency of these devices compare with a specified product.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Feng, Director, Principal Investigator — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China

REFERENCES:
- See also: Related Info — http://www.zsph.com/